CLINICAL TRIAL: NCT04880278
Title: Multimodal Assessment of Cannabinoid Target Engagement in Adults With Obsessive-Compulsive Disorder
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Principal Investigator is no longer at the Institution and a request for early termination of the grant supporting the study was submitted to NIH.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7809; K23MH125315 (NIH)
Record Dates: First submitted 2021-04-29; First posted 2021-05-10 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Nabilone; Fear Extinction; Threat Response; Goal-directed vs. Habitual Behavior; fMRI
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nabilone (Active Comparator): In a randomized, double-blind, placebo-controlled design, we will administer a one-time oral dose of nabilone (1mg) or placebo approximately two hours prior to fMRI scanning and task performance in 60 adults with OCD.
  Interventions: Drug: Nabilone
- Placebo (Placebo Comparator): In a randomized, double-blind, placebo-controlled design, we will administer a one-time oral dose of nabilone (1mg) or placebo approximately two hours prior to fMRI scanning and task performance in 60 adults with OCD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Half of the participants (30 individuals) will receive nabilone 1mg. Nabilone will be placed in opaque capsules with dextrose filler and administered by mouth only once (around 120 minutes prior to fMRI scanning).
  Other Names: Cesamet (brand name)
  Arms: Nabilone
Drug: Placebo — Half of the participants (30 individuals) will receive placebo capsules that are opaque and contain only dextrose. Placebo capsules will be administered by mouth only once (around 120 minutes prior to fMRI scanning).
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test how a medication called nabilone (Cesamet) affects neurocognitive processes involved in obsessive-compulsive disorder (OCD), including threat response, processing of fear signals, and habitual behavior. OCD is a disabling illness that affects around 2% of the population and involves recurrent intrusive thoughts (obsessions) and repetitive behaviors (compulsions) that lead to distress and/or impaired functioning. Nabilone is a synthetic form of delta-9-tetrahydrocannabinol (THC, the primary psychoactive component of the cannabis plant). It acts on the brain's endocannabinoid system, which has been hypothesized to play a role in OCD symptoms. Nabilone is approved by the FDA for the treatment of chemotherapy-induced nausea and vomiting. It is not FDA-approved for treating OCD.

In this study, 60 adults with OCD will receive a single dose of either nabilone or placebo. Participants will then complete a series of assessments including neuroimaging, psychophysiology (e.g., skin conductance recording), computerized behavioral tasks, and self-report measures. The information gained from this study could contribute to the development of new treatments for people with OCD and related disorders.

DETAILED DESCRIPTION:
The total time required for each participant is 4 visits, as outlined below:

Visit 1: Screening, Questionnaires, and Orientation: During this visit potential participants will learn about the study procedures, sign the informed consent documents, complete diagnostic evaluations and medical screening with study staff. Participants will also complete a series of forms that ask about demographic information, OCD symptoms, use of drugs and alcohol, and other aspects of physical and mental health.

Visit 2: Behavioral Tests: During this visit participants will complete several computer tasks. Study staff will measure reaction time and obtain psychophysiological information (e.g., skin conductance recordings). The tasks that the participant completes will involve viewing images within a virtual environment. An aversive stimulus (e.g., loud burst of noise, animated snake) may follow one image most of the time, while other images may never be followed by a noise or a snake. The participant will need to try to predict whether the aversive cue will occur or not based on which image is shown, and will be asked to repeatedly rate on a scale how likely they think it is that a noise/snake will occur after each image.

Visit 3: Behavioral Tests with Drug or Placebo and MRI scan: For safety reasons, participants will be asked not to take any drugs for at least 24 hours before this visit. They will also be asked not to use marijuana/cannabis for at least 2 weeks before participating. Participants will be required to test negative on a urine drug screen and breathalyzer before continuing with this visit; women must also have a negative pregnancy test. Participants will need to complete a field sobriety test at the end of this visit and will be asked not to drive or operate machinery for the following 24 hours; participants not traveling to the clinic by subway or taxi should arrange to have a friend or family member pick them up.

Two hours before beginning the Visit 3 tasks, participants will be asked to swallow a capsule containing either nabilone or placebo (sugar pill). Nabilone is a Food & Drug Administration (FDA) approved medication, and the dose (1mg, one time) is unlikely to have any effects that last beyond the duration of the study visit. About every 30 minutes after taking the pill, the participant will fill out some questionnaires asking about how they are feeling at the moment. At the end of the session, they will also be asked to guess whether they received nabilone or placebo.

Participants will then complete a task that is similar to the one on the previous day (Visit 2), but will be completed in the MRI scanner. During the MRI scan, participants will view the same images as on the previous day (Visit 2), and may experience the same aversive stimulus as during Visit 2. They will again be asked to rate how much they expect to experience the aversive stimulus after each image and to self-report their level of anxiety on a scale from 0 to 100. Finally, they will be asked to relax with their eyes open while viewing a white fixation cross on a back background.

Participants will complete an additional task outside of the MRI scanner. Participants will be repeatedly asked to view and choose between different images (e.g., spaceships), which lead to a different set of images. They must select one image from this second set, with some choices leading to a small monetary reward.

Visit 4: Behavioral Tests and MRI scan: This visit will be very similar to Visit 3, except that participants will not receive any study medication. Participants will complete the same type of task inside the MRI scanner, while the study staff measures reaction time, psychophysiological response, and brain activation. Participants will view the same images as in Visits 2 and 3, and may experience the same aversive stimulus. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and to report their level of anxiety on a scale from 0 to 100. Participants will again be asked to relax with their eyes open while viewing a white fixation cross on a black background. Finally, outside of the scanner, participants will complete another decision-making task similar to the one they completed the day before.

ELIGIBILITY:
Inclusion Criteria:

* Between 21-55 years of age
* Physically healthy and, if female, not pregnant
* Able to tolerate all study procedures
* Able to provide written informed consent to participate
* Right-handed
* Primary diagnosis of OCD
* Not taking psychotropic medications or other substances likely to interact with nabilone

Exclusion Criteria:

* History of any significant medical condition that may increase the risk of participation
* Females who are pregnant or nursing
* Current or lifetime history of psychiatric disorders other than OCD that may increase the risk of participation (e.g. lifetime psychosis or bipolar disorder)
* Current substance use disorder
* Positive urine toxicology or alcohol breathalyzer
* Any history of adverse reaction to a cannabinoid
* History of receiving cognitive behavior or exposure-based psychotherapy in the past 3 months
* History of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
* History of claustrophobia or unable to tolerate confined spaces like an MRI

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Brain Measure 1 | 5 years
  Functional magnetic resonance imaging (fMRI) BOLD percent signal change within regions of interest (e.g., amygdala; ventromedial prefrontal cortex; hippocampus) during task performance
Brain Measure 2 | 5 years
  Difference in fMRI resting state functional connectivity
Skin conductance response (SCR) | 5 years
  Change in SCR (peak amplitude from 0.5-4.5 sec following stimulus presentation minus average 2 second baseline prior to stimulus presentation).
Electromyography (EMG) | 5 years
  Change in orbicularis oculi EMG response (peak-to-peak value in the 21-150ms after stimulus presentation)
Expectancy Ratings | 5 years
  To assess the expected likelihood that an aversive cue (e.g. noise burst or animated snake) will occur or not based on which image was shown, participants will repeatedly rate their expectancy of the aversive cue using a button box on a scale from 1 to 3 (1 = certain that the aversive cue will be presented; 2 = certain that the aversive cue will not be presented; 3 = uncertain whether the aversive cue will be presented).

SECONDARY OUTCOMES:
Two-step task performance | 5 years
  Computational modeling will be applied to examine the balance between model-free vs. model-based behavior based on the relative frequency of outcomes selected at each stage of the task (i.e., Choice 1 vs. Choice 2).
Subjective Units of Distress | 5 years
  Subjective Units of Distress (SUDS): Self-reported fear/anxiety on a scale from 0-100; taken at three time points throughout the tasks: before the task begins, in the middle of the task, and at the end of the task.
Yale-Brown Obsessive-Compulsive Challenge Scale | Collected on Visit 3, immediately before capsule ingestion (Time 0), and 30, 60, 120, 180, and 240 minutes afterwards.
  Measure of self-reported obsessions and compulsions over short timeframes (e.g., minutes to hours).
Spielberger State/Trait Anxiety Inventory (STAI) | Collected on Visit 3, immediately before capsule ingestion (Time 0), and 30, 60, 120, 180, and 240 minutes afterwards.
  Self-report measure of trait anxiety and of current anxiety symptoms
Visual Analog Scales (VAS) | Collected on Visit 3, immediately before capsule ingestion (Time 0), and 30, 60, 120, 180, and 240 minutes afterwards.
  Measures self-report of current OCD and anxiety symptoms on a visual scale of 1-10
Nabilone Side Effects Checklist | Collected on Visit 3, immediately before capsule ingestion (Time 0), and 30, 60, 120, 180, and 240 minutes afterwards.
  Self-report checklist of potential nabilone side effects on a scale of 1-4 (absent, mild, moderate, severe)
Drug Effects Questionnaire (DEQ) | Collected on Visit 3, immediately before capsule ingestion (Time 0), and 30, 60, 90, 120, 150, 180, and 240 minutes afterwards, as well as at 8 hours and 24 hours afterwards.
  Self-report measure of intoxicating effects on a scale of 1-4
End of Session Questionnaire (ESQ) | 5 years
  A brief questionnaire that asks participants about their experiences during the experimental session
Heart rate | Heart rate will be collected at the following intervals during Visit 3: Immediately before capsule ingestion (Time 0), and 30, 60, 120, 180, and 240 minutes afterwards.
  Heart rate in beats per minute
Blood pressure | Blood pressure will be collected at the following intervals during Visit 3: Immediately before capsule ingestion (Time 0), and 30, 60, 120, 180, and 240 minutes afterwards.
  Blood pressure (systolic blood pressure/diastolic blood pressure; units: mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Reilly Kayser, MD, Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No